CLINICAL TRIAL: NCT06679348
Title: Comparison of Physiological Responses of Virtual Reality Walking Exercise Compared to Walking Performed on Treadmills in Healthy Individuals
Brief Title: Exploring Physiological Responses of Virtual Reality Walking Exercise Versus Treadmill Walking in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, SOzkan, asst.prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Autonomous Nervous System
Record Dates: First submitted 2024-11-01; First posted 2024-11-07 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-10

CONDITIONS: Autonomous Nervous System; Fatigue
Keywords: treadmill; virtual reality; heart rate variability; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Walking Exercise (Experimental): Walking in virtual reality combined with treadmill exercise
  Interventions: Other: Treadmill walking exercise using VR
- Walking on Treadmill (Experimental): walking on treadmills
  Interventions: Other: walking exercise on treadmill

INTERVENTIONS:
Other: walking exercise on treadmill — The study included two intervention groups, consisting of participants who met the inclusion criteria and adhered to the experimental procedures. One group will do treadmill walking exercises, while the other will do treadmill walking exercises using virtual reality (VR). Both interventions were conducted in a single session, with each group participating in a 20-minute walking exercise session at a moderate intensity, as identified by other studies.
  Arms: Walking on Treadmill
Other: Treadmill walking exercise using VR — Walking on the treadmill with the Free Run game on the Nintendo Wii allows users to walk at 5 miles per hour for 20 minutes. The user gets on the Wii Balance Board and starts walking in the virtual environment after running the application. The application detects the user's movements and controls the progress of the virtual character. During this experience, users increase their motivation by encountering various landscapes while tracking their performance and getting information about the calories they spend. This setup provides a fun, game-like atmosphere for a realistic walking experience.
  Arms: Virtual Reality Walking Exercise

SUMMARY:
This study aimed to systematically compare the physiological responses generated by walking exercises conducted in a VR environment versus those performed on a treadmill, with a specific focus on their impacts on the autonomic nervous system and fatigue levels

DETAILED DESCRIPTION:
This study was designed as a single-blind, randomized controlled trial. It was conducted in accordance with the Declaration of Helsinki, adhering to ethical principles for medical research involving human participants. Faculty of health sciences students from İstanbul Atlas University were invited to participate in this study. The inclusion criteria were as follows: aged between 18 and 25 years; classified as inactive or minimally active according to the International Physical Activity Questionnaire score; voluntary consent to participate; and a body mass index (BMI) of ≤30 kg/m².

Participants were excluded from the study if they met any of the following conditions: presence of visual, auditory, vestibular, or neurological deficits; a history of inflammatory diseases, surgeries, or cancer; any cardiopulmonary disorders, including asthma, within the last six months; major musculoskeletal injuries sustained within the last six months; other health issues that could compromise safety during exercise; or conditions known to affect autonomic nervous system (ANS) function, such as diabetes mellitus or autonomic neuropathy or current smoking status or failure to adhere to the experimental procedures of our study.

Our study comprehensively examines the effects of virtual reality (VR) walking exercise and traditional treadmill walking on autonomic nervous system (ANS) and fatigue levels during recovery.

Investigations into the physiological responses elicited by VR exercise interventions underscore a critical gap in our understanding of how VR modalities produce distinct responses compared with conventional exercise forms, particularly treadmill walking.

ELIGIBILITY:
Inclusion Criteria:

* classified as inactive or minimally active according to the International Physical Activity Questionnaire score
* voluntary consent to participate
* body mass index (BMI) of ≤30 kg/m²

Exclusion Criteria:

* presence of visual, auditory, vestibular, or neurological deficits
* a history of inflammatory diseases, surgeries, or cancer
* any cardiopulmonary disorders, including asthma, within the last six months
* major musculoskeletal injuries sustained within the last six months
* function, such as diabetes mellitus or autonomic neuropathy
* current smoking status

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
autonomic nervous system and fatigue levels | Assessments were conducted at four key time points: before the exercise session (T1), immediately after exercise completion (T2), and during the recovery phase at ten minutes post-exercise (T3) and thirty minutes post-exercise (T4).
  1. Autonomic Nervous System Function
     Measure: Heart Rate Variability (HRV) via Polar H10 chest strap. Unit of Measure: Milliseconds (ms) for HRV, reflecting autonomic balance. Interpretation: Higher HRV scores typically indicate better autonomic nervous system regulation, suggesting increased vagal tone and resilience to stress.
  2. Fatigue Levels
  Measure: OMNI Scale of Perceived Exertion (OMNI). Unit of Measure: OMNI Scale ranges from 0 (no fatigue) to 10 (maximum fatigue). Interpretation: Higher scores indicate greater perceived exertion and fatigue, while lower scores suggest less perceived exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Kagıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes